CLINICAL TRIAL: NCT06479213
Title: REACH (Restore Energy, Activity Can Help) Lupus Study
Acronym: REACH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00004759; K23AR078177 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-06-28 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-04

CONDITIONS: Systemic Lupus Erythematosus; Fatigue
Keywords: Physical activity; Peer coaching; Mobile health application; Chronic disease self-management
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Fatigue; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REACH Peer Coaching Program (Experimental): Participants will receive access to the REACH mobile health application and a REACH peer coach with whom they will meet weekly during the 12 weeks of the program.
  Interventions: Behavioral: REACH Peer Coaching Program; Behavioral: REACH Mobile Health Application
- REACH Mobile Health Application (Active Comparator): Participants will receive access to the REACH mobile health application which they will use during the 12 weeks of the program.
  Interventions: Behavioral: REACH Mobile Health Application

INTERVENTIONS:
Behavioral: REACH Peer Coaching Program — The REACH Peer Coaching Program consists of weekly coaching calls conducted over video teleconference. Coaches will use motivational interviewing to help participants formulate and work towards movement goals.
  Arms: REACH Peer Coaching Program
Behavioral: REACH Mobile Health Application — Participants will use the the REACH mobile health application to set weekly movement goals and log physical activity.

SUMMARY:
The goal of this clinical trial is to pilot test the REACH peer coaching program for fatigue in people with systemic lupus erythematosus. The main questions it aims to answer are:

1. Is the REACH program feasible and acceptable to participants?
2. What is the impact of the REACH program on fatigue?

Researchers will compare the REACH peer coaching program to the REACH mobile health application to see if the REACH program works to reduce fatigue.

Participants will:

* Use the REACH mobile health application to set weekly movement goals and log daily physical activity
* Meet weekly with their REACH peer coach (if they have one) to talk about their movement goals and progress
* Complete weekly symptom surveys
* Complete study surveys when they start the program, in the middle of the program, at the end of the program, and 12 weeks after the program ends
* Participate in an interview to provide feedback on the program

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic lupus erythematosus based on 2019 American College of Rheumatology classification criteria
* ≥ 18 years of age
* English-speaking
* Ownership of a smartphone
* Physician's permission to participate in the study (including engagement in physical activity)
* Fatigue Severity Scale score ≥ 4

Exclusion Criteria:

* Inability to consent or comply with the study protocol (cognitively impaired adults).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 6 months
  Enrollment rates (subjects enrolled/eligible individuals approached).
Adherence | 12 months
  Proportions of educational modules, activity logs, and coaching sessions completed.
Acceptability | 12 to 24 weeks
  Net Promoter Scores for the educational modules, REACH app, and REACH peer coaching intervention. Interviews exploring the acceptability of study procedures (e.g. data collection methods, study assessments, functionality of the mobile app) and engagement with educational modules and peer coaches.

SECONDARY OUTCOMES:
Fatigue | 12 weeks and 24 weeks
  Effect size estimate of change in fatigue using the Fatigue Severity Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gulati N, Singh K, Morrissey E, Calvache P, Rose-Smith J, Gore-Massy M, Chiu F, Trinquart L, Navarro-Millan I, Folta S, Kasturi S. Study protocol for a randomized controlled trial to pilot Restore Energy, Activity Can Help (REACH): an mHealth-enabled peer coaching intervention for fatigue in systemic lupus erythematosus. Contemp Clin Trials Commun. 2025 Jun 7;46:101508. doi: 10.1016/j.conctc.2025.101508. eCollection 2025 Aug. PMID 40548142
- See also: Study Landing Page — https://redcap.link/REACH_Study